CLINICAL TRIAL: NCT00697502
Title: A Phase I Study of Capecitabine In Patients With Solid Tumors
Brief Title: Study of Capecitabine In Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Haematology-Oncology, Dr. Ross Soo, National University Hospital, Singapore
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PG03/32/06
Record Dates: First submitted 2008-06-11; First posted 2008-06-16 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Solid Tumors
MeSH Terms: interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 2: TSER 3R/3R (Experimental): Cohorts of 3-6 patients in each genotype group will receive escalating doses of capecitabine until MTD is reached. Once MTD is determined, an additional 6-9 patients (for a total of 12 patients) will receive treatment at that dose.
  Interventions: Drug: Capecitabine
- Group 1: TSER 2R/2R or 2R/3R (Experimental): Cohorts of 3-6 patients in this genotype group will receive escalating doses of capecitabine until MTD is reached. Once MTD is determined, an additional 6-9 patients (for a total of 12 patients) will receive treatment at that dose.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine — Capecitabine (XELODA) is supplied as biconvex, oblong film-coated tablets for oral administration and will be obtained from NUH Cancer Centre pharmacy.
  Each light peach-colored tablet contains 150 mg capecitabine and each peach-colored tablet contains 500 mg capecitabine. Capecitabine is to be administered orally within 30 minutes after the end of a meal (breakfast, dinner). Tablets should be swallowed with about 200 mL of water (not fruit juices). Capecitabine will be administered for 14 days followed by a 7 day rest period.
  Other Names: XELODA

SUMMARY:
Hypothesis:

Patients with TYMS 2R/2R or 2R/3R appear to be more sensitive to fluoropyrimidines, conferring a higher risk of grade 3-4 fluoropyrimidine related toxicity and a higher response rate compared with 3R/3R. The genotype 3R/3R is more common in East Asia and is associated with greater tolerability to fluoropyrimidine as measured by lower toxicity but also lower response rates. As sensitivity to fluoropyrimidine appears to be affected by TYMS genotype, we hypothesise that patients with TYMS 3R/3R are more tolerant to standard doses of capecitabine and require higher doses to overcome fluoropyrimidine resistance. We designed this study to develop TYMS genotype specific dosing of capecitabine.

Aims:

1. To determine the maximal tolerated dose (MTD) of capecitabine twice a day for two weeks followed by one week rest period (intermittent schedule) in patients with the advanced/ and or metastatic cancer based on TYMS genotype.
2. To determine a suitable phase II dose of intermittent schedule capecitabine.
3. To determine the safety and toxicity of this regimen.
4. To perform plasma pharmacokinetics of capecitabine.
5. To determine the relationship between genes of relevance in the fluoropyrimidine pathway with pharmacokinetics and toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Cytologically or histologically confirmed advanced or metastatic non- hematologic malignancy that had failed previous therapies or cancer for which there are no standard treatment options.
2. Presence of at least one uni-dimensional measurable lesion as defined by the RECIST criteria.
3. Required genotype characteristics:

   * Group 1: TSER genotype 2R/2R or 2R/3R
   * Group 2: TSER genotype 3R/3R
4. Able to swallow capsules
5. Age>=18 years
6. Kanorfsky performance status of at least 70% or ECOG performance status <2 (Appendix A)
7. Life expectancy of at least 3 months
8. Hb >=9 g/dL
9. ANC >=1.5 x 10^9/L
10. Platelet count >=100 x 10^9/L.
11. Total bilirubin and serum creatinine <=1.5x upper limits of normal reference range (ULN)
12. Alkaline phosphatase, AST/ALT levels <=2.5x upper limit of normal. If hepatic metastases are present, these parameters could be <=10x the ULN.
13. Women of reproductive age and men must agree to practice effective contraception during the entire study period. Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-child- bearing potential. Females with childbearing potential must have a negative serum pregnancy test within 7days prior to study enrolment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
14. Signed written informed consent

Exclusion Criteria:

1. Received any anti-cancer therapy including chemotherapy, immunotherapy, radiotherapy, hormonal, biologic or any investigational therapy within 28 days prior to study drug administration (6 weeks for mitomycin or nitroureas) and not recovered.
2. Patients who have not recovered from major surgery
3. Any woman pregnant or lactating.
4. Known CNS metastases
5. Renal impairment with a creatinine clearance <=50mL/min (as calculated according to Cockcroft and Gault formula) or serum creatinine > ULN
6. Clinically significant cardiac disease, eg. Congestive cardiac failure, symptomatic coronary heart disease, cardiac arrhythmia or myocardial infarction within the last 12 months.
7. Known HIV infection
8. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, other serious uncontrolled concomitant disease, psychiatric illness/ social situation that would limit study compliance.
9. Known allergies to any component of the study drug
10. Lack of physical integrity of the upper gastrointestinal tract or those with malabsorption syndrome
11. Organ allografts
12. Known dihydropyrimidine dehydrogenase deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
To determine the maximal tolerated dose (MTD) of capecitabine twice a day for two weeks followed by one week rest period (intermittent schedule) in patients with the advanced/ and or metastatic cancer based on TYMS genotype. | 4 weeks

SECONDARY OUTCOMES:
Plasma concentrations of capecitabine and its metabolites | 3 weeks
  Pharmacokinetic sampling will be performed during cycle 1 on days 1 and 14 at the following time points:
  Baseline (predose), and 15 min, 30 min, 1 hr, 2 hr, 4 hr, 5 hr and 6 hr after dosing. Blood samples will be centrifuged at 1500 g and 4oC for 10 min and supernatant plasma removed and stored below -20oC until analysis. Plasma concentrations of capecitabine and its metabolites will be quantified by a validated liquid chromatography with mass-spectrometry detection (LC-MS-MS) method

CONTACTS AND LOCATIONS:
Overall Officials: Ross Andrew Soo, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Soong R, Diasio RB. Advances and challenges in fluoropyrimidine pharmacogenomics and pharmacogenetics. Pharmacogenomics. 2005 Dec;6(8):835-47. doi: 10.2217/14622416.6.8.835. PMID 16296946
- [Background] Park DJ, Stoehlmacher J, Zhang W, Tsao-Wei D, Groshen S, Lenz HJ. Thymidylate synthase gene polymorphism predicts response to capecitabine in advanced colorectal cancer. Int J Colorectal Dis. 2002 Jan;17(1):46-9. doi: 10.1007/s003840100358. PMID 12018454